CLINICAL TRIAL: NCT00107627
Title: Skin Incision Study - Closure of Skin Incisions in Gynecological Cancer Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Responsible Party: Professor Andreas Obermair, Queensland Centre for Gynaecological Cancer
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SIS001
Record Dates: First submitted 2005-04-06; First posted 2005-04-07 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Cancer
Keywords: Gynaecological Cancer; Surgical Staples; Subcuticular Sutures
MeSH Terms: conditions — Neoplasms | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Skin staples;
  Interventions: Other: Skin staples;
- 2 (Active Comparator): Monocryl subcuticular sutures.
  Interventions: Other: Monocryl subcuticular sutures.
- 3 (Active Comparator): Caprosyn subcuticular sutures.
  Interventions: Other: Caprosyn subcuticular sutures.

INTERVENTIONS:
Other: Caprosyn subcuticular sutures. — Caprosyn subcuticular sutures.
  Other Names: Sutures; Stitches
  Arms: 3
Other: Monocryl subcuticular sutures. — Monocryl subcuticular sutures.
  Other Names: Sutures,; Stitches
  Arms: 2
Other: Skin staples; — Skin staples;
  Other Names: Staples
  Arms: 1

SUMMARY:
The Skin Incision Study evaluates the efficacy of skin closure methods: skin staples and subcuticular sutures at 6 weeks and at 3 months following the operation by measuring cosmesis and pain.

DETAILED DESCRIPTION:
The Surgical Skin Incisions (SSI) is an investigator initiated, randomized, prospective (pilot) study comparing methods of skin closure following gynecological cancer surgery to evaluate:

* cosmesis;
* pain;
* adverse events.

The two most common methods of skin incision closure are staples or subcuticular sutures. Adverse events to surgical incisions represent major and significant burdens to patients and the health care system; however, no data is available comparing methods of skin closure. Surgeons have traditionally had to use personal belief rather than data or evidence to choose the method of skin incision closure. This study evaluates three types of skin closure methods:

* Skin staples;
* Monocryl subcuticular sutures;
* Caprosyn subcuticular sutures.

The objective of this trial is to evaluate the efficacy of sutures and staples at 6 weeks and at 3 months following the operation by measuring cosmesis and pain. These are assessed by both the patient and the surgeon independently using linear analogue scales and by collecting information on analgesic medications taken by the patient. The safety of the staples and sutures will be expressed by the incidence of adverse events following surgery. Post-operative events such as wound infection, other wound complications, grade of inflammation, hemorrhage and other complications will be graded according to the Common Toxicity Criteria (CTC version 3) and recorded.

Investigators will invite public patients with proven or suspected gynecological cancer from Royal Brisbane and Women's Hospital and Mater Hospital (RBWH) that are booked to have elective surgery and that meet the selection criteria to participate in this study.

This is a pilot study to generate data for a definitive randomized study. Ninety (90) patients are required for recruitment to the pilot study.

The type of closure method patients will receive will be allocated using a randomization process. Three equally sized study arms of 30 patients will have their surgical incision closed with either surgical staples, Monocryl or Caprosyn. Additionally, patients will be stratified by site so as to remove selection bias.

All tests and assessments before and after the operation are standard of care. These results will be recorded. No additional tests or assessments will be performed for the aim of this trial.

Randomization, data management and statistical analysis will be coordinated by the Queensland Centre for Gynaecological Cancer. Statistical analysis will include calculating mean values and standard deviations for scores for each group at each assessment. Chi-square tests will be used to compare differences in proportions of patients who did or did not experience adverse events at each time point.

Results of this trial will be presented at scientific meetings at a national and international level and at educational meetings with medical staff. The results of this trial will also be submitted for publishing. The study will generate data for a definitive randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Public patients at RBWH and at the Mater Public Hospital booked for elective surgery (laparotomy)
* Surgery for suspected or proven gynecological cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient compliance and geographic proximity that allow adequate follow-up
* Signed written informed consent
* Females >=18 years of age

Exclusion Criteria:

* Unplanned laparotomy
* Laparoscopic procedures
* Unwillingness of the patient to participate in the trial
* Non-compliance of participant
* Unavailability for follow-up
* Patients who are unable or unwilling to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of the device as measured by cosmesis, pain and requirement for analgesic and antibiotic medication | 6 weeks after surgery

SECONDARY OUTCOMES:
To evaluate the wound healing process (normal or delayed), cosmesis and pain, requirement for surgical or medical intervention (analgesic and antibiotic medication) | 3 months after surgery
Safety of the device as expressed in the incidence of adverse events following surgery | 6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Principal Investigator — Queensland Centre for Gynaecological Cancer
Locations (2):
- Australia (2):
  - QCGC, Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Public Hospital, South Brisbane, Queensland